CLINICAL TRIAL: NCT04757376
Title: A Double-blind, Randomized, Active-controlled, Phase 3 Study to Compare Efficacy, Pharmacokinetics, Pharmacodynamics, and Safety of CT-P41 and US-licensed Prolia in Postmenopausal Women With Osteoporosis
Brief Title: A Phase 3 Study to Compare Between CT-P41 and US-licensed Prolia in Postmenopausal Women With Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P41 3.1; 2020-005974-91 (EudraCT Number)
Record Dates: First submitted 2021-02-12; First posted 2021-02-17 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-05

CONDITIONS: Postmenopausal Women With Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CT-P41 (Experimental): 60 mg/mL single dose administration, Solution for injection in prefilled syringe(PFS)
  Interventions: Biological: CT-P41
- US-licensed Prolia (Active Comparator): 60 mg/mL single dose administration, Solution for injection in PFS
  Interventions: Biological: US-licensed Prolia

INTERVENTIONS:
Biological: CT-P41 — 60 mg/mL single dose, Solution for injection in PFS
  Arms: CT-P41
Biological: US-licensed Prolia — 60 mg/mL single dose, Solution for injection in PFS
  Arms: US-licensed Prolia

SUMMARY:
This study is a Double-blind, Randomized, Active-controlled, Phase 3 Study to Compare Efficacy, Pharmacokinetics, Pharmacodynamics, and Safety of CT-P41 and US-licensed Prolia in Postmenopausal Women with Osteoporosis

DETAILED DESCRIPTION:
This is a double-blind, randomized, active-controlled, Phase 3 study to evaluate the efficacy, PK, PD, and safety including immunogenicity of CT-P41 compared with US-licensed Prolia in postmenopausal women with osteoporosis. All patients will also receive daily supplementation containing at least 1,000 mg of elemental calcium and at least 400 IU vitamin D from randomization to EOS visit and the data will be collected via patient's diary.

ELIGIBILITY:
Inclusion Criteria:

1. Women, 50 to 80 years of age, both inclusive.
2. Body weight between 40.0 and 99.9 kg, both inclusive, when rounded to the nearest tenth.
3. Postmenopausal
4. Bone mineral density T-score ≤ - 2.5 and ≥ - 4.0 at the lumbar spine (L1 to L4) as assessed by the central imaging vendor based on dual-energy X-ray absorptiometry(DXA) scan.
5. Patients must have at least 3 vertebrae considered evaluable at the lumbar spine (L1 to L4) and at least 1 hip considered evaluable by DXA scan assessed by the central imaging vendor. Patients with unilateral metal in hips that would be allowed for the other side of 1 evaluable hip are included.
6. Patient with albumin-adjusted total serum calcium ≥ 8.5 mg/dL (≥ 2.125 mmol/L) at Screening.

Exclusion Criteria:

1. Patient previously received denosumab, any other monoclonal antibodies, or biologic agents for osteoporosis
2. Patient confirmed or suspected with infection of COVID-19 at Screening, or has contact with COVID-19 patient within 14 days from Screening
3. Patient with history and/or presence of one severe or > 2 moderate vertebral fractures as determined by central reading of lateral spine X-ray
4. Patient with history and/or presence of hip fracture
5. Patient with history and/or presence of hyperparathyroidism or hypoparathyroidism, irrespective of current controlled or uncontrolled status
6. Patient with current hyperthyroidism (unless well controlled on stable antithyroid therapy)
7. Patient with current hypothyroidism (unless well controlled on stable thyroid replacement therapy)
8. Patient with history and/or presence of bone disease and metabolic disease (except for osteoporosis) that may interfere with the interpretation of the results

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 479 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-11-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- Estonia (4):
  - Center For Clinical And Basic Research, Tallinn, Harju
  - East Tallinn Central Hospital-Ravi 18, Tallinn, Harju
  - Clinical Research Centre Ltd, Tartu, Tartu
  - KLV Arstikabinet, Pärnu
- Latvia (2):
  - Health Center Association, Medical Center Liepaja, Liepāja
  - Health Center 4-117 K. Barona Str, Riga
- Poland (10):
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Poznaniu, Poznan, Greater Poland Voivodeship
  - Centrum Medyczne Poznan - PRATIA - PPDS, Skórzewo, Greater Poland Voivodeship
  - Krakowskie Centrum Medyczne, Krakow, Lesser Poland Voivodeship
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial we Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - SOMED CR Sp. z o.o. Sp. Komandytowa - Lodz, Lódz, Lódzkie
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw, Masovian Voivodeship
  - SOMED CR Sp. z o.o. Sp. Komandytowa - Warszawa, Warsaw, Masovian Voivodeship
  - NZOZ Osteo Medic SC Artur Racewicz Jerzy Supronik, Bialystok, Podlaskie Voivodeship
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia, Pomeranian Voivodeship
  - MCM Krakow - PRATIA - PPDS, Krakow
- Ukraine (4):
  - AES - AS - Medical Center of Edelweiss Medics LLC, Kyiv
  - Clinic of SI Institute of Gerontology n.a. D.F.Chebotaryov of NAMS of Ukraine, Kyiv
  - AES - AS - Medical Center of Medbud - Clinic LLC, Kyiv
  - Clinic of SRI of Invalid Rehab. (ESTC) of VNMU n.a. M.I.Pyrohov, Vinnytsia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment was conducted in 20 study centers in 4 countries.
Pre-assignment Details: The screening period began after the participants had signed the written informed consent form and completed it within 28 days before the 1st randomization (Week 0 Day 1). On Week 0 Day 1, participants were randomized in a 1:1 ratio to receive CT-P41 or US-Prolia during Treatment Period (TP) I. At Week 52 predose, participants in the US-Prolia group were re-randomized 1:1 to either continue US-Prolia or transition to CT-P41. The participants in the CT-P41 group continued with CT-P41 for TP II.
Groups:
- CT-P41: A total of 2 subcutaneous administration of 60 mg CT-P41 (proposed denosumab biosimilar) at Week 0 and Week 26 (26-week intervals) in TP I
  CT-P41: 60 mg/mL single dose, Solution for injection in PFS
- US-licensed Prolia: A total of 2 subcutaneous administration of 60 mg US-licensed Prolia (denosumab) at Week 0 and Week 26 (26-week intervals) in TP I
  US-licensed Prolia: 60 mg/mL single dose, Solution for injection in PFS
- CT-P41 Maintenance: Participants treated with CT-P41 in TP I continued the treatment with CT-P41 as a third dose at Week 52 in TP II
- US-licensed Prolia Maintenance: Participants treated with US-Prolia in TP I were re-randomized to continue the treatment with US-licensed Prolia as a third dose at Week 52 in TP II
- Switched to CT-P41: Participants treated with US-licensed Prolia in TP I were re-randomized to switch to CT-P41 as a third dose at Week 52 in TP II
Period: TP I - Week 0, Day 1 to Week 52 Predose
Arm/Group | CT-P41 | US-licensed Prolia | CT-P41 Maintenance | US-licensed Prolia Maintenance | Switched to CT-P41
Started | 240 | 239 | 0 | 0 | 0
Completed (completed the study treatment in TP I) | 221 | 201 | 0 | 0 | 0
Not Completed | 19 | 38 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 24 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 5 | 0 | 0 | 0
Not completed — Protocol Violation | 5 | 4 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 3 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Disease progression | 0 | 1 | 0 | 0 | 0
Not completed — Terminated the study before the initiation of the study treatment | 1 | 1 | 0 | 0 | 0
Period: TP II - Week 52 to Week 78
Arm/Group | CT-P41 | US-licensed Prolia | CT-P41 Maintenance | US-licensed Prolia Maintenance | Switched to CT-P41
Started | 0 | 0 | 221 | 100 | 101
Completed (completed the study treatment in TP II) | 0 | 0 | 220 | 100 | 101
Not Completed | 0 | 0 | 1 | 0 | 0
Not completed — Discontinued the study treatment before the study treatment initiation due to the adverse event | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The overall number of participants analyzed represents the Intent-to-treat (ITT) Set. The ITT set was defined as all participants randomly assigned to receive study drug (CT-P41 or US-Prolia), regardless of whether or not any study drug was administered.
Groups:
- Total: Total of all reporting groups
Arm/Group | CT-P41 | US-licensed Prolia | Total
Number analyzed (Participants) | 240 | 239 | 479
Age, Continuous [Median (Full Range); unit: years] | 66.0 [50 to 79] | 66.0 [51 to 79] | 66.0 [50 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 240 | 239 | 479
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race - White | 240 | 239 | 479
  Ethnicity - Hispanic or Latino | 0 | 3 | 3
  Ethnicity - Non-Hispanic or Non-Latino | 240 | 236 | 476
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 24.92 (4.230) | 25.23 (4.328) | 25.08 (4.277)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mineral Density (BMD) at Week 52 - Full Analysis Set (FAS)
Description: Bone mineral density was assessed by dual-energy X-ray absorptiometry (DXA) and assessments of the lumbar spine (L1 to L4) were performed at a central imaging vendor. To evaluate the difference between 2 groups in the primary efficacy endpoint, the percent change from baseline in BMD for lumbar spine (L1 to L4) by DXA at Week 52 was analyzed using an analysis of covariance (ANCOVA) model coupled with multiple imputation assuming the data to be missing at random (MAR).
Time Frame: baseline (screening), Week 52 predose
Population: The FAS was defined as all participants who received at least 1 full dose of the study drug (CT-P41 or US-licensed Prolia). The total number of participants in FAS was 239 and 238 in the CT-P41 and US-licensed Prolia groups, respectively. The overall number of participants analyzed represents the number of participants in FAS who had a BMD assessment result for the lumbar spine by DXA at Week 52.
Measure: Least Squares Mean (Standard Error); unit: percentage change (%)
Arm/Group | CT-P41 | US-licensed Prolia
Number analyzed (Participants) | 222 | 212
percentage change (%) | 4.9597 (0.29977) | 5.1528 (0.32133)
Statistical Analysis 1: Comparison: CT-P41 vs US-licensed Prolia; Test type: Equivalence — Statistical equivalence: the 90% confidence interval (CI) of the difference in the mean of the primary efficacy endpoint between treatment groups was entirely within an equivalence margin, [- 1.45, + 1.45]; ANCOVA; ANCOVA included the treatment as a fixed effect and age, baseline LS-BMD T-score, and prior bisphosphonates therapy (Yes versus No) as covariates; Mean Difference (Final Values) = -0.19, 90% CI 2-sided [-0.76 to 0.38]

2. Secondary Outcome: Percent Change From Baseline in Lumbar Spine, Total Hip, and Femoral Neck BMD at Week 52 - FAS
Description: Bone mineral density was assessed by DXA and assessments of the lumbar spine (L1 to L4), total hip, and femoral neck were performed at a central imaging vendor.
Time Frame: baseline (screening), Week 52 predose
Population: The overall number of participants analyzed row represents the total number of participants in the FAS. The number analyzed per row represents the number of participants in FAS with lumbar spine, total hip, or femoral neck BMD value at baseline and Week 52.
Measure: Mean (Standard Deviation); unit: percentage change (%)
Arm/Group | CT-P41 | US-licensed Prolia
Number analyzed (Participants) | 239 | 238
percentage change (%)
  Lumbar spine: number analyzed (Participants) | 222 | 212
  Lumbar spine | 5.4913 (3.79907) | 5.6621 (3.75768)
  Total hip: number analyzed (Participants) | 219 | 212
  Total hip | 2.7914 (2.87044) | 2.4253 (2.84061)
  Femoral neck: number analyzed (Participants) | 219 | 212
  Femoral neck | 2.2295 (4.02031) | 1.9476 (3.86739)

3. Secondary Outcome: Percent Change From Baseline in Lumbar Spine, Total Hip, and Femoral Neck BMD at Week 78 - FAS-TP II Subset
Description: Bone mineral density was assessed by DXA and assessments of the lumbar spine (L1 to L4), total hip, and femoral neck BMD were performed at a central imaging vendor.
Time Frame: baseline (screening), Week 78
Population: The FAS-TP II subset was defined as all participants in FAS who received 1 full dose of the study drug (CT-P41 or US-licensed Prolia) at Week 52. The overall number of participants analyzed row represents the total number of participants in the FAS-TP II subset. The number analyzed per row represents the number of participants in FAS-TP II subset with lumbar spine, total hip, or femoral neck BMD value at baseline and Week 78.
Measure: Mean (Standard Deviation); unit: percentage change (%)
Arm/Group | CT-P41 Maintenance | US-licensed Prolia Maintenance | Switched to CT-P41
Number analyzed (Participants) | 220 | 100 | 101
percentage change (%)
  Lumbar spine: number analyzed (Participants) | 213 | 97 | 98
  Lumbar spine | 6.8588 (4.12795) | 6.5745 (3.40437) | 7.0532 (3.55985)
  Total hip: number analyzed (Participants) | 213 | 96 | 98
  Total hip | 3.4706 (2.81017) | 2.7947 (2.79862) | 3.3837 (2.92786)
  Femoral neck: number analyzed (Participants) | 213 | 96 | 98
  Femoral neck | 2.9995 (3.73072) | 2.4429 (3.61786) | 2.8226 (4.02021)

4. Secondary Outcome: Incidence of New Vertebral, Nonvertebral, and Hip Fractures During TP I - FAS
Description: Efficacy analysis of new vertebral fractures included only vertebral fractures occurring from T4 to L4 and confirmed by the central imaging vendor. A new vertebral fracture was defined as an increase of ≥1 grade in any vertebra from T4 to L4 that was normal at screening.
  The nonvertebral fractures endpoint included fractures other than those of the vertebrae, excluding the skull, facial bones, mandible, metacarpals, and phalanges (fingers or toes) since they are not associated with decreased BMD, and excluded pathologic fractures and those associated with severe trauma acquired from a fall (from a height higher than a stool, chair, or first rung of a ladder) or otherwise. Only nonvertebral fractures confirmed by the central imaging vendor were included in the efficacy analysis.
  The fractures occurring at the site of femur neck, femur intertrochanter, or femur subtrochanter were considered as a hip fracture.
Time Frame: up to Week 52 predose
Population: The overall number of participants analyzed and the number analyzed represents the total number of participants in FAS.
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P41 | US-licensed Prolia
Number analyzed (Participants) | 239 | 238
Participants
  New vertebral fracture | 1 | 1
  Nonvertebral fracture | 2 | 4
  Hip fracture | 0 | 0

5. Secondary Outcome: Incidence of New Vertebral, Nonvertebral, and Hip Fractures During TP II - FAS-TP II Subset
Description: as for outcome 4
Time Frame: from Week 52 to Week 78
Population: The overall number of participants analyzed and the number analyzed represents the total number of participants in FAS-TP II subset.
Measure: Count of Participants; unit: Participants
Groups:
- US-licensed Prolia Maintenance: Participants treated with US-licensed Prolia in TP I were re-randomized to continue the treatment with US-licensed Prolia as a third dose at Week 52 in TP II
Arm/Group | CT-P41 Maintenance | US-licensed Prolia Maintenance | Switched to CT-P41
Number analyzed (Participants) | 220 | 100 | 101
Participants
  New vertebral fracture | 1 | 0 | 0
  Nonvertebral fracture | 2 | 0 | 1
  Hip fracture | 0 | 0 | 0

6. Secondary Outcome: Trough Serum Concentration (Ctrough) of Denosumab at Weeks 0 and 26 - Pharmacokinetic (PK) Set
Description: The Ctrough, a concentration before the next study drug administration, was calculated by non-compartmental analysis method from the concentration-time data. All serum concentrations below the lower limit of quantification (LLoQ) was set to 0 in the descriptive summaries of PK parameter estimation. In TP I, the Ctrough of denosumab at Weeks 0 and 26 was assessed as the serum concentration at Weeks 26 and 52 before the study drug administration, respectively.
Time Frame: Week 0 Day 1 predose, Week 26 predose
Population: The PK Set was defined as all participants who received at least 1 full dose of the study drug (CT-P41 or US-licensed Prolia) and had at least 1 post-treatment PK concentration data with a concentration above the LLoQ prior to dosing at Week 52. The overall number of participants analyzed row represents the total number of participants in PK Set. The number analyzed per row represents the number of participants in PK set with data at the corresponding time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CT-P41 | US-licensed Prolia
Number analyzed (Participants) | 237 | 236
ng/mL
  Week 0 Day 1: number analyzed (Participants) | 227 | 221
  Week 0 Day 1 | 46.79 (105.102) | 31.69 (73.253)
  Week 26: number analyzed (Participants) | 221 | 207
  Week 26 | 75.64 (154.630) | 63.99 (140.912)

7. Secondary Outcome: Ctrough of Denosumab at Week 52 - PK-TP II Subset
Description: The Ctrough, a concentration before the next study drug administration, was calculated by non-compartmental analysis method from the concentration-time data. All serum concentrations below the LLoQ was set to 0 in the descriptive summaries of PK parameter estimation. In TP II, the Ctrough of denosumab at Week 52 was assessed as the serum concentration at Week 78.
Time Frame: Week 52
Population: The PK-TP II subset was defined as all participants in the PK set who received 1 full dose of the study drug (CT-P41 or US-licensed Prolia) at Week 52 and had at least 1 post-treatment PK concentration data with a concentration above the LLoQ after Week 52. The overall number of participants analyzed row represents the number of participants in the PK-TP II subset who had the Ctrough data at Week 52.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CT-P41 Maintenance | US-licensed Prolia Maintenance | Switched to CT-P41
Number analyzed (Participants) | 214 | 96 | 98
ng/mL | 70.24 (126.852) | 66.60 (129.573) | 126.15 (508.689)

8. Secondary Outcome: Maximum Serum Concentration (Cmax) of Denosumab After First Dose - PK Set
Description: Cmax was calculated by non-compartmental analysis method from the concentration-time data. All serum concentrations below the LLoQ was set to 0 in the descriptive summaries of PK parameter estimation.
Time Frame: from baseline (Week 0 Day 1 predose) to Week 26 predose
Population: Participants in the PK Set who had assessments of Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | CT-P41 | US-licensed Prolia
Number analyzed (Participants) | 237 | 236
ng/mL | 5851.2 (32.2) | 5492.7 (29.8)

9. Secondary Outcome: Percent Change From Baseline for Serum Concentration of Serum Carboxy-terminal Cross-linking Telopeptide of Type I Collagen (s-CTX) at Weeks 26 and 52 - Pharmacodynamic (PD) Set
Description: Serum concentration below the LLoQ was set to the LLoQ. The percent change from baseline for serum concentration at each visit was calculated as ([Result at each visit - Result at Baseline] / Result at Baseline) × 100.
Time Frame: Baseline (Week 0 Day 1 predose), Weeks 26 and 52 (predose)
Population: The PD set was defined as all participants who received a full dose of the study drug (CT-P41 or US-licensed Prolia) at Day 1 (Week 0) and had at least 1 post-treatment PD concentration data with a concentration above the LLoQ before dosing at Week 52. The overall number of participants analyzed represents the total number of participants in PD set. The number analyzed per row represents the number of participants in the PD set who had the data at the corresponding time point.
Measure: Median (Inter-Quartile Range); unit: percentage change (%)
Arm/Group | CT-P41 | US-licensed Prolia
Number analyzed (Participants) | 237 | 236
percentage change (%)
  Week 26: number analyzed (Participants) | 227 | 220
  Week 26 | -75.6972 [-83.7838 to -59.8504] | -74.3547 [-81.8667 to -63.0572]
  Week 52: number analyzed (Participants) | 221 | 207
  Week 52 | -72.7506 [-85.8306 to -57.1429] | -72.5275 [-82.8794 to -56.6188]

10. Secondary Outcome: Percent Change From Baseline for Serum Concentration of s-CTX at Week 78 - PD-TP II Subset
Description: as for outcome 9
Time Frame: Baseline (Week 0 Day 1 predose), Week 78
Population: The PD-TP II subset was defined as all participants in the PD set who received 1 full dose of the study drug (CT-P41 or US-licensed Prolia) at Week 52 and had at least 1 post-treatment PD concentration data with a concentration above the LLoQ after Week 52. The overall number of participants analyzed represents the number of participants in the PD-TP II subset who had s-CTX value at baseline and Week 78.
Measure: Median (Inter-Quartile Range); unit: percentage change (%)
Arm/Group | CT-P41 Maintenance | US-licensed Prolia Maintenance | Switched to CT-P41
Number analyzed (Participants) | 214 | 97 | 98
percentage change (%) | -70.4609 [-81.0680 to -46.4052] | -64.9063 [-78.9644 to -48.6034] | -70.1268 [-84.3162 to -47.4940]

11. Secondary Outcome: Percent Change From Baseline for Serum Concentration of Procollagen Type 1 N-terminal Propeptide (P1NP) at Weeks 26 and 52 - PD Set
Description: as for outcome 9
Time Frame: Baseline (Week 0 Day 1 predose), Weeks 26 and 52 (predose)
Population: The overall number of participants analyzed represents the total number of participants in PD Set. The number analyzed per row represents the number of participants in PD set who had P1NP value at the corresponding time point.
Measure: Median (Inter-Quartile Range); unit: percentage change (%)
Arm/Group | CT-P41 | US-licensed Prolia
Number analyzed (Participants) | 237 | 236
percentage change (%)
  Week 26: number analyzed (Participants) | 226 | 221
  Week 26 | -69.31 [-76.69 to -57.78] | -68.22 [-76.79 to -56.68]
  Week 52: number analyzed (Participants) | 220 | 207
  Week 52 | -69.99 [-76.77 to -50.26] | -66.61 [-76.56 to -53.16]

12. Secondary Outcome: Percent Change From Baseline for Serum Concentration of P1NP at Week 78 - PD-TP II Subset
Description: Serum concentration below the LLoQ was set to the LLoQ. The percent change from baseline for serum concentration was calculated as ([Result at each visit - Result at Baseline] / Result at Baseline) × 100.
Time Frame: Baseline (Week 0 Day 1 predose), Week 78
Population: The overall number of participants analyzed represents the number of participants in the PD-TP II subset who had the P1NP value at baseline and Week 78.
Measure: Median (Inter-Quartile Range); unit: percentage change (%)
Arm/Group | CT-P41 Maintenance | US-licensed Prolia Maintenance | Switched to CT-P41
Number analyzed (Participants) | 214 | 97 | 98
percentage change (%) | -67.05 [-76.20 to -53.24] | -68.60 [-75.12 to -50.11] | -64.54 [-78.00 to -53.92]

13. Secondary Outcome: Number of Participants With at Least 1 Anti-drug Antibodies (ADA)/Neutralizing Antibodies (NAb) Result After the First Study Drug Administration of TP I - Safety Set
Description: Samples that were positive in the ADA confirmatory assay were analyzed further to conduct a NAb assessment. The test outcomes for the screening assay were 'Positive' or 'Negative'. The number of patients with at least one ADA/NAb positive result after the first study drug administration of each treatment period including scheduled and unscheduled visits (Treatment Period I: Week 0 / Treatment Period II: Week 52) regardless of their ADA status at baseline were presented.
Time Frame: up to Week 52 predose
Population: The Safety set was defined as all participants who received at least 1 dose (full or partial) of the study drug (CT-P41 or US-licensed Prolia). The overall number of participants analyzed and the number analyzed represents the total number of participants in the Safety Set.
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P41 | US-licensed Prolia
Number analyzed (Participants) | 239 | 238
Participants
  ADA positive | 233 | 234
  NAb positive | 0 | 0

14. Secondary Outcome: Number of Participants With at Least 1 ADA/NAb Result After the First Study Drug Administration of TP II - Safety-TP II Subset
Description: as for outcome 13
Time Frame: from Week 52 to Week 78
Population: The Safety-TP II subset was defined as all participants in the Safety set who received 1 dose (full or partial) of study drug (CT-P41 or US-licensed Prolia) at Week 52. The overall number of participants analyzed and the number analyzed represents the number of participants in the Safety-TP II subset.
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P41 Maintenance | US-licensed Prolia Maintenance | Switched to CT-P41
Number analyzed (Participants) | 220 | 100 | 101
Participants
  ADA positive | 208 | 92 | 93
  NAb positive | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Through Week 78 - Treatment Period I: Adverse event start date before the study drug administration in Treatment Period II - Treatment Period II: Adverse event start date on or after the date of study drug administration in Treatment Period II.
Description: Among the 240 in the CT-P41 group and 239 in the US-licensed Prolia group who initiated Treatment Period I, one participant each terminated the study participation before the first study treatment administration.
  Since the adverse events results in Treatment Period I was summarized in the safety set who received at least 1 dose of the study drug during Treatment Period I, the total number of participants at risk was 239 and 238 in the CT-P41 and US-licensed Prolia groups, respectively.
Arm/Group | CT-P41 | US-licensed Prolia | CT-P41 Maintenance | US-licensed Prolia Maintenance | Switched to CT-P41
All-Cause Mortality (participants affected / at risk) | 1/239 | 0/238 | 1/220 | 0/100 | 0/101
Serious Adverse Events (participants affected / at risk) | 7/239 | 10/238 | 8/220 | 3/100 | 0/101
Other Adverse Events (participants affected / at risk) | 98/239 | 86/238 | 44/220 | 14/100 | 29/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CT-P41 (N=239) | US-licensed Prolia (N=238) | CT-P41 Maintenance (N=220) | US-licensed Prolia Maintenance (N=100) | Switched to CT-P41 (N=101)
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Hormone level abnormal (Investigations) | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Borderline ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Genital neoplasm malignant female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Vulval leukoplakia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CT-P41 (N=239) | US-licensed Prolia (N=238) | CT-P41 Maintenance (N=220) | US-licensed Prolia Maintenance (N=100) | Switched to CT-P41 (N=101)
COVID-19 (Infections and infestations) | 28 | 26 | 8 | 3 | 6
Upper respiratory tract infection (Infections and infestations) | 25 | 20 | 13 | 4 | 11
Urinary tract infection (Infections and infestations) | 12 | 4 | 6 | 0 | 3
Nasopharyngitis (Infections and infestations) | 10 | 12 | 4 | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 21 | 7 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 | 13 | 2 | 1 | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 15 | 5 | 6 | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-04-18): https://cdn.clinicaltrials.gov/large-docs/76/NCT04757376/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-10): https://cdn.clinicaltrials.gov/large-docs/76/NCT04757376/SAP_001.pdf